CLINICAL TRIAL: NCT06329375
Title: Food Insecurity Reduction & Strategy Team
Acronym: FIRST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Neera Ahuja, Professor of Medicine, Associate Chief Medical Officer- Inpatient Care Services, Division Chief- Hospital Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 72967
Record Dates: First submitted 2024-02-29; First posted 2024-03-25 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2; Food Insecurity; Diabetes Mellitus, Type 1
Keywords: inpatient
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1 | interventions — Food Assistance

STUDY DESIGN:
Intervention Model Description: Participants will be prospectively randomized into either a nutrition program (intervention), or receiving state-of-the-art standard of care (SOC) in a 4:1 ratio. Patients in the intervention group will be provided the following two resources in addition to SOC:
  1. Enhanced access to nutritious food (twice daily meal delivery up to 90 days post-discharge),
  2. Education at discharge and continuing outreach to enhance knowledge for better diet and food options
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SoC group (No Intervention): Standard of care (SOC)
- Nutrition program (Intervention) (Experimental): Patients in the intervention group will be provided the following two resources in addition to SOC:
  1. Enhanced access to nutritious food (twice daily meal delivery up to 90 days post-discharge).
  2. Education at discharge and continuing outreach to enhance knowledge for better diet and food options.
  Interventions: Other: Nutrition program

INTERVENTIONS:
Other: Nutrition program — Nutrition program with twice daily meal delivery up to 90 days post-discharge and food and diet education at discharge.
  Arms: Nutrition program (Intervention)

SUMMARY:
This study seeks to address the multifaceted challenges posed by food disparities and their negative consequences on health outcomes, via a comprehensive community health intervention program. Study objectives include:

1. To describe the social-demographic and clinical factors associated with food insecurity in the hospitalized diabetic population.
2. To design, implement and evaluate a nutrition program targeting the hospitalized diabetic population. The investigators will prospectively randomize the target population into either a nutrition program (Intervention), or state-of-art standard of care (SOC) in a 4:1 ratio. Participants in the intervention group will be provided the following two resources in addition to SOC: 1) Enhanced access to nutritious food (twice daily meal delivery up to 90 days post-discharge) 2) Education at discharge and continuing outreach to enhance knowledge for better diet and food options.
3. To enhance community engagement and develop a systematic implementation plan for long-term roll-out of the nutrition program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1 or Type 2 Diabetes Mellitus
* Admitted to Stanford Healthcare inpatient unit
* Residence in California at time of enrollment
* Positive Screening for Food Insecurity
* On a Healthcare Plan covered by Mom's Meals.

Exclusion Criteria:

* Plans to be discharged to a skilled nursing facility.
* Patients who prefer a language for which a short-form consent is not available.
* No Home Address
* Pregnant Participants.
* No access to refrigerator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Food insecurity at 60 -days post initial discharge | 60 days from discharge
  Primary outcome is whether the participant had food insecurity in the past 30 days, measured at 60-days post initial discharge by the Food Insecurity Reduction and Strategy Team (FIRST) Survey Instrument questionnaire.
  1. Within the past 30 days, you were worried that your food would run out before you got the money to buy more. (Categorical)
     a. Never true, Sometimes true, Often true, Patient refused
  2. Within the past 30 days, the food you bought just didn't last and you didn't have money to get more. (Categorical)
     1. Never true, Sometimes true, Often true, Patient refused

SECONDARY OUTCOMES:
Food insecurity at 30- and 90- days post post initial discharge | 30-, and 90- days from discharge
  The secondary outcome is whether the participant had food insecurity in the past 30 days, measured at 30-days and 90-days post initial discharge by the Food Insecurity Reduction and Strategy Team (FIRST) Survey Instrument questionnaire:
  1. Within the past 30 days, you were worried that your food would run out before you got the money to buy more. (Categorical)
     a. Never true, Sometimes true, Often true, Patient refused
  2. Within the past 30 days, the food you bought just didn't last and you didn't have money to get more. (Categorical)
     1. Never true, Sometimes true, Often true, Patient refused
Measures of diabetes stress | 30-,60-, and 90- days from discharge
  Feeling overwhelmed by the demands of living with Diabetes measured using ordinal scale with range 1-6.
Measures of hypoglycemia | 30-,60-, and 90- days from discharge
  Whether ever having a low blood sugar (low glucose or hypoglycemic) reaction in the past 4 weeks and number of times having a low blood sugar (low glucose or hypoglycemic) reaction in the past 4 weeks. (ordinal scale: 0, 1-3, 4-7, 8+)
Measures of medication adherence | 30-,60-, and 90- days from discharge
  Proportion of participants who missed their recommended diabetes medication in the past 7 days at least once and the mean number of days that the medication was missed in the past 7 days, measured using measured by participant self-report during survey response collection at 30-,60-, and 90-days post-discharge.
Hospitalization | 30-,60-, and 90- days from discharge
  Proportion of participants having overnight hospitalizations in the past 30 days and mean number of nights with overnight hospitalizations in the past 30 days measured by participant self-report during survey response collection at 30-,60-, and 90-days post-discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Neera Ahuja, MD, Principal Investigator — Stanford University; Christine Santiago, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Medicine, Palo Alto, California, United States